CLINICAL TRIAL: NCT05576532
Title: The Efficacy and Safety of Venetoclax Plus IM2 Regimen for Relapsed and Refractory T Lymphoblastic Lymphoma/Leukemia
Brief Title: Venetoclax Plus IM2 Regimen for Relapsed and Refractory T Lymphoblastic Lymphoma/Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, principal investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHXYXY-2022-VEN-T-LBL
Record Dates: First submitted 2022-10-09; First posted 2022-10-12 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: T-lymphoblastic Lymphoma; Relapsed Disease; Refractory Lymphoma; Refractory Leukemia; Safety; Efficacy, Self
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bcl-2 inhibitor plus IM2 regimen (Experimental): bcl-2 inhibitor plus IM2 regimen
  Interventions: Drug: BCL2 Inhibitor plus IM2 regimen

INTERVENTIONS:
Drug: BCL2 Inhibitor plus IM2 regimen — oral bcl-2 inhibitor plus IM2(Ifosfamide plus Mitoxantrone or Idarubicin plus methotrexate) chemotherapy

SUMMARY:
To evaluate the safety and efficacy of Venetoclax plus IM2 regimen for relapsed and refractory T lymphoblastic lymphoma/leukemia. Dosage of Venetoclax:100mg/d-400mg/d(dose adjustment when concomitant used with CYP3A inhibitor) for 1-28 days (at least 7 days); IM2 regimen: Ifosfamide 1-1.5g/m2/d for 5 days; Mitoxantrone 6-8g/m2/d for 3 days( or Liposome mitoxantrone 20mg/m2 d1 or Idarubicin 6-8mg/m2/d for 3 days) ;methotrexate 1-1.5g/m2/d for 1 day;

ELIGIBILITY:
Inclusion Criteria

Fourteen to 45 Years Old, Male and female; Expected survival > 12 weeks; ECOG score 0-2; Confirmed diagnosis of T lymphoblastic lymphoma： a. Patients who do not get a PR with ≥2 induction chemotherapy or a CR with ≥ 4 induction chemotherapy b. Relapsed patients c. For any Patients who failed ASCT/allo-SCT d.The disease can be assessed (BM or CT scan) Confirmed diagnosis of acute T lymphoblastic leukemia (disease involved in BM, and no signs of lymph nodes or mass involvement): Patients who do not get a CR with ≥2 prior induction therapy such as Hyper-A and B regimens. b. relapsed after CR with chemotherapy c. For any Patients failed ASCT/allo-SCT Liver, kidney, and cardiopulmonary functions meet the following requirements: a. Ccr≥60mL/min(Cockcroft Gault) b. Left ventricular ejection fraction >50%; c.Baseline oxygen saturation>92%; d. Total bilirubin ≤ 1.5×ULN; e. ALT and AST≤ 3×ULN; Able to understand and sign the Informed Consent

Exclusion Criteria:

Malignant tumors other than T cell malignancies within 5 years prior to screening, in addition, to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection; Uncontrolled infection including bacterial or virus or fungal disease; patients with positive HBsAg or HBcAb and positive peripheral blood HBV DNA titer detection; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; syphilis positive; Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease; Any uncontrolled disease may affect entry Current or history of CNS involvement by malignancy.Known history or presence of clinically relevant central nervous system (CNS) pathology.Patients with a known history or prior diagnosis of other immunologic or inflammatory disease affecting the CNS (such as epilepsy) Pregnant or lactating woman, and a female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion; Active or uncontrollable infection requiring systemic therapy Known be allergic to Venetoclax or Ifosfamide or Mitoxantrone or Idarubicin or methotrexate The investigators consider other conditions unsuitable for enrollment. Early relapse(time from the end of IM2 regimen to relapse within 6 months ) post- or refractory to IM2 chemotherapy Patients who may not be able to sign the Informed Consent due to disease,or who do not understand or unwillingness or inability to comply with research requirements

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate after 2 cycles of chemotherapy | 2 months after chemotherapy
  complete response rate plus partial response rate
Overall response rate after 4 cycles of chemotherapy | 4 months after chemotherapy
  complete response rate plus partial response rate
Grade 3-4 Adverse events incidence | 28 days after chemotherapy
  Grade 3-4 Adverse events incidence

SECONDARY OUTCOMES:
Overall survival | 12 months
  OS for patients enrolled
Progression free survival | 12 months
  PFS for patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin G Song, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China